CLINICAL TRIAL: NCT05739214
Title: The Effect of Combined Red and Infrared Lasers on Histopathology Collagen Formation in Diabetic Foot Ulcer: a Randomized Controlled Trial
Brief Title: The Effect of Combined Red and Infrared Lasers on Histopathology Collagen Formation in Diabetic Foot Ulcer
Acronym: wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heidy F. Ahmed, Doctor of physical therapy certified wound specialist at Al kasr Al Anini teaching hospital, Cairo, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NILES-EC-CU 23/3/3
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Diabetic Foot; Wound Heal; Collagen Diseases
Keywords: infrared laser; red laser; chronic diabetic foot ulcer; collagen formation
MeSH Terms: conditions — Diabetic Foot; Collagen Diseases | interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: group A received laser therapy in sequential mode, group B received laser therapy in separate mode and the control group C receive conventional wound care treatment
Who Masked: Participant, Outcomes Assessor
Masking Description: the patient didn't know the types of modes of laser applied even in the control group i used light not laser to equalize the blindness
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- laser sequential mode (Experimental): All patients received 2 sessions of laser therapy / week with different wavelengths in sequential mode in two consecutive months of treatment aiming complete wound closure , patients received & infrared laser therapy plus traditional wound care
  Interventions: Device: laser therapy
- laser seperate mode (Experimental): All patients received 2 sessions of laser therapy / week with different wavelengths in seperate mode in two consecutive months of treatment aiming complete wound closure , patients received & infrared laser therapy plus traditional wound care
  Interventions: Device: laser therapy
- traditional wound care (Active Comparator): Traditional wound care inform of
  1. Wound care treatment
     * Debridement to remove necrotic tissue
     * Irrigation of the wound by normal saline
     * Change dressing daily to protect wound from infection
  2. Foot care
     * Wash feet daily, dry carefully especially between toe
     * Avoid extreme temperatures
     * Inspection daily of foot blisters
  3. Foot wear
     * Avoid walking bare foot
     * Properly fitted shoes
     * Avoid wearing open-toed shoes
  Interventions: Device: laser therapy

INTERVENTIONS:
Device: laser therapy — All patients received 2 sessions of laser therapy / week in two consecutive months of treatment aiming complete wound closure , patients received & infrared laser therapy plus traditional wound care:
  (I) Use red & infrared laser therapy device with 4 different wavelengths in a synchronized mode:
  1. 980 nm for wound decontamination, improve circulation, lymphatic drainage
  2. 915 nm enhances O2 delivery
  3. 810 nm increases ATP production
  4. 650 nm accelerate surface healing, tissue regeneration plus traditional wound treatment mentioned before

SUMMARY:
Objective: investigate The effect of combined red and infrared lasers on histopathology collagen formation in diabetic foot ulcer Participants: The forty five patients will assigned randomly into three equal groups, each group consist of 15 patients, group A received laser therapy in sequential mode, group B received laser therapy in separate mode and the control group C receive conventional wound care treatment

DETAILED DESCRIPTION:
Objective: investigate The effect of combined red and infrared lasers on histopathology collagen formation in diabetic foot ulcer Participants: The forty five patients will assigned randomly into three equal groups, each group consist of 15 patients, group A received laser therapy in sequential mode, group B received laser therapy in separate mode and the control group C receive traditional wound care Outcomes: the primary outcomes were the wound surface area measurement, % of wound complete closure and % of collage formation before and after receiving the treatment protocol for two consequetive months

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 60 years; both gender; Diabetic patients type II; Ulcer lasting longer than two months; diabetic foot ulcer (DFU) grade 1 (Superficial diabetic ulcer, ulcer limited to the dermis, not extending to the subcutis) or grade 2 (Ulcer of the skin extending through the subcutis with exposed tendon or bone and without osteomyelitis or abscess formation) according to the Wagner classification

Exclusion Criteria:

* Patients with fixed ankle deformity as Charcot foot or stiffness; Patients with any type of osteomyelitis associated with DFU; the presence of active infection requiring hospitalization, gangrene, systemic diseases such as collagen-vascular diseases, renal failure, evidence of ischemia; BMI < 30 kg/m2 as Obesity can cause poor perfusion due to vascular insufficiencies; an altered population of immune mediators may lengthen the inflammatory process & decrease oxygenation of subcutaneous adipose tissue which is liable to be infected

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
percent of collagen formation | two consecutive months
  by histological pictures
percent of wound size measurement methods | two consecutive months
  measure percent of wounds decrease surface area

SECONDARY OUTCOMES:
percent of wounds complete closure | two consecutive months
  measure percent of wounds complete closure in each group

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S El Basiouny, professor, Principal Investigator — national institute of laser sciences; Heidy F Ahmed, master, Principal Investigator — Kasr al aini
Locations (1):
- Al Kasr Al Aini Teaching Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD), all IPD that underline results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: In the next month of registration.
Access Criteria: Information will be available upon request through the following e-mail: heidy.fouad@gmail.com.

REFERENCES:
- [Background] Hegazi R, El-Gamal M, Abdel-Hady N, Hamdy O. Epidemiology of and Risk Factors for Type 2 Diabetes in Egypt. Ann Glob Health. 2015 Nov-Dec;81(6):814-20. doi: 10.1016/j.aogh.2015.12.011. PMID 27108148
- [Background] Banik PC, Barua L, Moniruzzaman M, Mondal R, Zaman F, Ali L. Risk of diabetic foot ulcer and its associated factors among Bangladeshi subjects: a multicentric cross-sectional study. BMJ Open. 2020 Feb 28;10(2):e034058. doi: 10.1136/bmjopen-2019-034058. PMID 32114471
- [Background] American Diabetes Association. Peripheral arterial disease in people with diabetes. Diabetes Care. 2003 Dec;26(12):3333-41. doi: 10.2337/diacare.26.12.3333. No abstract available. PMID 14633825
- [Background] Vinik AI, Erbas T, Park TS, Nolan R, Pittenger GL. Platelet dysfunction in type 2 diabetes. Diabetes Care. 2001 Aug;24(8):1476-85. doi: 10.2337/diacare.24.8.1476. PMID 11473089
- [Background] Sorensen MLB, Jansen RB, Wilbek Fabricius T, Jorgensen B, Svendsen OL. Healing of Diabetic Foot Ulcers in Patients Treated at the Copenhagen Wound Healing Center in 1999/2000 and in 2011/2012. J Diabetes Res. 2019 Sep 8;2019:6429575. doi: 10.1155/2019/6429575. eCollection 2019. PMID 31583251
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2009 Jan;32 Suppl 1(Suppl 1):S62-7. doi: 10.2337/dc09-S062. No abstract available. PMID 19118289
- [Background] Cunha JLS, Carvalho FMA, Pereira Filho RN, Ribeiro MAG, de Albuquerque-Junior RLC. Effects of Different Protocols of Low-Level Laser Therapy on Collagen Deposition in Wound Healing. Braz Dent J. 2019 Jul 22;30(4):317-324. doi: 10.1590/0103-6440201902400. PMID 31340220
- [Background] 8) Brandão, M. G. S. A., Ximenes, M. A. M., de Oliveira Ramalho, A., Veras, V. S., Barros, L. M., & de Araújo, T. M. (2020). Effects of low-level laser therapy on the healing of foot ulcers in people with diabetes mellitus. Estima-Brazilian Journal of Enterostomal Therapy, 18, e320.
- [Background] Oyebode O, Houreld NN, Abrahamse H. Photobiomodulation in diabetic wound healing: A review of red and near-infrared wavelength applications. Cell Biochem Funct. 2021 Jul;39(5):596-612. doi: 10.1002/cbf.3629. Epub 2021 Apr 18. PMID 33870502
- [Background] Coerper S, Wicke C, Pfeffer F, Koveker G, Becker HD. Documentation of 7051 chronic wounds using a new computerized system within a network of wound care centers. Arch Surg. 2004 Mar;139(3):251-8. doi: 10.1001/archsurg.139.3.251. PMID 15006880
- [Background] Pierpont YN, Dinh TP, Salas RE, Johnson EL, Wright TG, Robson MC, Payne WG. Obesity and surgical wound healing: a current review. ISRN Obes. 2014 Feb 20;2014:638936. doi: 10.1155/2014/638936. eCollection 2014. PMID 24701367
- [Background] Kaviani A, Djavid GE, Ataie-Fashtami L, Fateh M, Ghodsi M, Salami M, Zand N, Kashef N, Larijani B. A randomized clinical trial on the effect of low-level laser therapy on chronic diabetic foot wound healing: a preliminary report. Photomed Laser Surg. 2011 Feb;29(2):109-14. doi: 10.1089/pho.2009.2680. Epub 2011 Jan 9. PMID 21214368
- [Background] Goralczyk K, Szymanska J, Szot K, Fisz J, Rosc D. Low-level laser irradiation effect on endothelial cells under conditions of hyperglycemia. Lasers Med Sci. 2016 Jul;31(5):825-31. doi: 10.1007/s10103-016-1880-4. Epub 2016 Feb 9. PMID 26861982
- [Background] Ayuk SM, Houreld NN, Abrahamse H. Collagen production in diabetic wounded fibroblasts in response to low-intensity laser irradiation at 660 nm. Diabetes Technol Ther. 2012 Dec;14(12):1110-7. doi: 10.1089/dia.2012.0125. Epub 2012 Oct 11. PMID 23057714
- [Background] Broughton G 2nd, Janis JE, Attinger CE. The basic science of wound healing. Plast Reconstr Surg. 2006 Jun;117(7 Suppl):12S-34S. doi: 10.1097/01.prs.0000225430.42531.c2. PMID 16799372
- [Background] Li S, Wang C, Wang B, Liu L, Tang L, Liu D, Yang G, Zhang L. Efficacy of low-level light therapy for treatment of diabetic foot ulcer: A systematic review and meta-analysis of randomized controlled trials. Diabetes Res Clin Pract. 2018 Sep;143:215-224. doi: 10.1016/j.diabres.2018.07.014. Epub 2018 Jul 23. PMID 30009935
- [Background] Morikawa M, Derynck R, Miyazono K. TGF-beta and the TGF-beta Family: Context-Dependent Roles in Cell and Tissue Physiology. Cold Spring Harb Perspect Biol. 2016 May 2;8(5):a021873. doi: 10.1101/cshperspect.a021873. PMID 27141051
- [Background] Huang J, Chen J, Xiong S, Huang J, Liu Z. The effect of low-level laser therapy on diabetic foot ulcers: A meta-analysis of randomised controlled trials. Int Wound J. 2021 Dec;18(6):763-776. doi: 10.1111/iwj.13577. Epub 2021 Mar 9. PMID 33751853